CLINICAL TRIAL: NCT05343130
Title: Efficacy of a Therapy With Brain-Computer Interface Controlled Functional Electrical Stimulation for Neurorehabilitation of Patients With Spinal Cord Injury (Eficacia de Una Terapia Con estimulación eléctrica Funcional Controlada Con Interfaz Cerebro-computadora Para neurorrehabilitación de Pacientes Con lesión Medular)
Brief Title: Efficacy of a Brain-Computer Interface Controlled Functional Electrical Stimulation Therapy for Spinal Cord Injury Neurorehabilitation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Nacional de Rehabilitacion (Other Government)
Collaborators: Instituto Tecnologico y de Estudios Superiores de Monterey (Other)
Responsible Party: Principal Investigator, Jessica Cantillo-Negrete, Researcher in Medical Sciences, Instituto Nacional de Rehabilitacion
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 10/22
Record Dates: First submitted 2022-04-18; First posted 2022-04-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Cervical Spinal Cord Injury
Keywords: brain-computer interface; functional electrical stimulation; motor rehabilitation; tetraplegia
MeSH Terms: conditions — Quadriplegia | interventions — Brain-Computer Interfaces

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Brain-Computer Interface controlled functional electrical stimulation feedback (Experimental)
  Interventions: Device: Brain-Computer Interface
- Sham Brain-Computer Interface controlled functional electrical stimulation feedback (Sham Comparator)
  Interventions: Device: Sham Brain-Computer Interface

INTERVENTIONS:
Device: Brain-Computer Interface — Hand movement will be elicited using functional electrical stimulation activated by the brain-computer interface based on hand movement intention.
  Arms: Brain-Computer Interface controlled functional electrical stimulation feedback
Device: Sham Brain-Computer Interface — Hand movement will be elicited using functional electrical stimulation which activation will be independent of the brain-computer interface based on hand movement intention.
  Arms: Sham Brain-Computer Interface controlled functional electrical stimulation feedback

SUMMARY:
The study's main goal is to determine the efficacy of a therapy with brain-computer interface controlled functional electrical stimulation for neurorehabilitation of spinal cord injury patients' upper limbs. For this purpose, a randomized controlled trial will be performed to compare the clinical and physiological effects of the brain-computer interface therapy with those of a sham intervention comprised by the application of functional electrical stimulation independently of brain-computer interface control.

ELIGIBILITY:
Inclusion Criteria:

* Spinal Cord Injury at neurological levels C6 or C7
* American Spinal Injury Association (ASIA) classification A, B, C or D
* Upper limb spasticity of less or equal to +1 measured with the Modified Ashworth Scale
* Time since disease onset of more than 6 months and less than 60 months
* Normal or corrected to normal vision

Exclusion Criteria:

* Severe attention deficits
* Previous diagnosis of traumatic brain injury
* Previous diagnosis of peripheral nerve injury
* Previous stroke diagnosis
* Previous diagnosis of neurodegenerative diseases
* History of fractures in upper extremities
* Skin lesions
* Contractures in upper extremities that hamper mobility
* Excessive muscle spasms

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Action Research Arm Test (ARAT) | At enrollment and after 7 weeks of the intervention onset
  Change of upper limbs function. Scale ranges from 0 to 57 points for each upper limb. A higher score means a better upper limb function.
Upper Extremity Motor Score (UEMS) | At enrollment and after 7 weeks of the intervention onset
  Change of upper limbs function. Scale ranges from 0 to 50 points if both upper limbs are assessed. A higher score means a better upper limb function.
Capabilities of Upper Extremities Questionnaire (CUE-Q) | At enrollment and after 7 weeks of the intervention onset
  Change of the functional limitation in tetraplegia. Scale ranges from 32 to 224 points if both upper limbs are assessed. A higher score means less functional limitation outcome.

SECONDARY OUTCOMES:
Spinal Cord Independence Measure III (SCIM-III) | At enrollment and after 7 weeks of the intervention onset
  Change of achievements of daily function. Scale ranges from 0 to 100 points. A higher score means a better capacity to perform activities of the daily living.
Life Satisfaction Questionnaire 9 (LISAT-9) | At enrollment and after 7 weeks of the intervention onset
  Change of life satisfaction. Scale ranges from 0 to 54 points. A higher score is expected with a better life satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Cantillo-Negrete, PhD, Principal Investigator — Instituto Nacional de Rehabilitacion (National Institute of Rehabilitation)
Locations (1):
- Instituto Nacional de Rehabilitacion Luis Guillermo Ibarra Ibarra (National Institute of Rehabilitation), Tlalpan, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data collected during the study will be available to other researchers from the principal investigator on reasonable request
Supporting Information: CSR
Time Frame: Six months after publication
Access Criteria: Researchers that make a request for access data and their request is approved by the National Institute of Rehabilitation Ethics Committee